CLINICAL TRIAL: NCT00636935
Title: Oral Corticosteroids Therapy and Interstitial Fibrosis in Patients With Pneumocystis Jirovecii Pneumonia (PCP) and pO2 of >70 at Presentation.
Brief Title: Corticosteroids Therapy and Pneumocystis Jirovecii Pneumonia (PCP)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient completed protocol
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Gary Simon, Principal Investigator, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARPCP001
Record Dates: First submitted 2008-02-28; First posted 2008-03-17 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pneumocystis Carinii Pneumonia
Keywords: Pneumocystis jirovecii Pneumonia; Corticosteroid Therapy; HIV; Pneumonia; Pulmonary Function Testing; Antibiotics; Prednisone; Human Immunodeficiency Virus; CD4; CD8; Viral Load; Bactrim; Pentamidine; Atovaquone; Primaquine/Clindamycin; Trimethoprim/Dapsone
MeSH Terms: conditions — Pneumonia, Pneumocystis; Pneumonia; Acquired Immunodeficiency Syndrome | interventions — Anti-Bacterial Agents; Adrenal Cortex Hormones; Prednisone; Trimethoprim, Sulfamethoxazole Drug Combination; Pentamidine; Atovaquone; Primaquine; Clindamycin; Trimethoprim; Dapsone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Antibiotic only therapy in patients with PCP and a pO2 of > 70mmHg.
  Interventions: Drug: Antibiotics only
- 2 (Experimental): Antibiotics and Corticosteroid therapy in patients with PCP and pO2 >70 mmHg.
  Interventions: Drug: Antibiotics + Corticosteroids
- 3 (Active Comparator): Standard of care therapy for patients with PCP and pO2 < 70mmHg.
  Interventions: Drug: Corticosteroids + antibiotics

INTERVENTIONS:
Drug: Antibiotics only — Antibiotic only for treatment for mild (pO2 > 70mmHg) PCP. Antibiotic Treatment with Bactrim, Pentamidine, Atovaquone, Primaquine/Clindamycin, or Trimethoprim/Dapsone.
  Arms: 1
Drug: Antibiotics + Corticosteroids — Prednisone 40mg orally twice daily for 11 days, followed by 40mg once daily for 5 days, followed by 20mg once daily for 5 days and antibiotics (Bactrim, Pentamidine, Atovaquone, Primaquine/Clindamycin, or Trimethoprim/Dapsone).
  Other Names: Prednisone; Bactrim; Pentamidine; Atovaquone; Primaquine/Clindamycin; Trimethoprim/Dapsone
  Arms: 2
Drug: Corticosteroids + antibiotics — Drugs will be prescribed per standard of care for patients with PCP and pO2 < 70mmHg.
  Other Names: Prednisone; Bactrim; Pentamidine; Atovaquone; Primaquine/Clindamycin; Trimethoprim/Dapsone
  Arms: 3

SUMMARY:
To explore the effects of corticosteroid therapy on pulmonary fibrosis and potentially pneumothorax in patients with mild PCP (pO2 >70mmHg) combined with the standard of care treatment of antibiotic therapy.

DETAILED DESCRIPTION:
Although the development of highly active anti-retroviral therapy has substantially reduced the incidence of Pneumocystis jirovecii pneumonia (PCP) among HIV-infected individuals, PCP remains one of the most common presenting opportunistic infection among this population. The use of adjunctive corticosteroids in the treatment of patients with moderate to severe PCP has resulted in a significant improvement in the development of respiratory failure and mortality.

Past studies have demonstrated no clinical benefit in patients with mild disease (pO2>75 torr on room air). This may have been due to the fact that few patients with mild disease develop either respiratory failure or die during the course of the acute illness so that a statistical difference could not be demonstrated.

However, considering parameters other than mortality, there is some evidence to suggest that patients with high pO2 concentrations benefit from adjunctive corticosteroids. PCP is associated with the development of pulmonary fibrosis and this can have significant consequences. Pathological studies have shown the development of interstitial fibrosis late in the course of acute illness. Studies have documented the presence of diffuse interstitial pneumonitis five months after the onset of acute illness. Therefore, patients with PCP infection, regardless of their pO2 level on presentation may benefit from corticosteroid therapy.

The current standard of care therapy for patients with PCP does not involve the addition of corticosteroids to standard antibiotics in those patients with pO2>70 mmHG. This study propose to conduct a randomized, prospective, un-blinded clinical trial to explore the effects of corticosteroid therapy on pulmonary fibrosis in patients with mild PCP who are admitted to the George Washington University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection,
* Hospital admission for suspected PCP,
* Confirmatory test for PCP (bronchoscopy with bronchoalveolar lavage), pO2>70 mmHg or pO2<70 mmHg while breathing room air,
* 18 years or older

Exclusion Criteria:

* Contraindications to corticosteroid therapy,
* Unable and or unwilling to perform PFTS or to return for follow-up evaluations,
* Underlying lung disease such as emphysema, untreated active tuberculosis, Uncontrolled diabetes (fasting glucose > 250 mg/dL,
* Uncontrolled hypertension (160/95 mmHg),
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary function testing and DLCO measurements in patients with PCP and pO2 > 70 mmHg. | 1 month, 3 months and 6 months after diagnosis
  Changes in pulmonary function testing and DLCO measurements in patients with PCP and pO2 > 70 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Afsoon Roberts, M.D., Principal Investigator — George Washington University Medical Faculty Associates
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozzette SA, Sattler FR, Chiu J, Wu AW, Gluckstein D, Kemper C, Bartok A, Niosi J, Abramson I, Coffman J, et al. A controlled trial of early adjunctive treatment with corticosteroids for Pneumocystis carinii pneumonia in the acquired immunodeficiency syndrome. California Collaborative Treatment Group. N Engl J Med. 1990 Nov 22;323(21):1451-7. doi: 10.1056/NEJM199011223232104. PMID 2233917
- [Background] Montaner JS, Lawson LM, Levitt N, Belzberg A, Schechter MT, Ruedy J. Corticosteroids prevent early deterioration in patients with moderately severe Pneumocystis carinii pneumonia and the acquired immunodeficiency syndrome (AIDS). Ann Intern Med. 1990 Jul 1;113(1):14-20. doi: 10.7326/0003-4819-113-1-14. PMID 2190515
- [Background] Nielsen TL, Eeftinck Schattenkerk JK, Jensen BN, Lundgren JD, Gerstoft J, van Steenwijk RP, Bentsen K, Frissen PH, Gaub J, Orholm M, et al. Adjunctive corticosteroid therapy for Pneumocystis carinii pneumonia in AIDS: a randomized European multicenter open label study. J Acquir Immune Defic Syndr (1988). 1992;5(7):726-31. PMID 1613673
- [Background] Gagnon S, Boota AM, Fischl MA, Baier H, Kirksey OW, La Voie L. Corticosteroids as adjunctive therapy for severe Pneumocystis carinii pneumonia in the acquired immunodeficiency syndrome. A double-blind, placebo-controlled trial. N Engl J Med. 1990 Nov 22;323(21):1444-50. doi: 10.1056/NEJM199011223232103. PMID 2233916
- [Background] Gallant JE, Chaisson RE, Moore RD. The effect of adjunctive corticosteroids for the treatment of Pneumocystis carinii pneumonia on mortality and subsequent complications. Chest. 1998 Nov;114(5):1258-63. doi: 10.1378/chest.114.5.1258. PMID 9823998
- [Background] Nowak J. Late pulmonary changes in the course of infection with Pneumocystis carinii. Acta Med Pol. 1966;7(1):23-41. No abstract available. PMID 5296368
- [Background] Whitcomb ME, Schwarz MI, Charles MA, Larson PH. Interstitial fibrosis after Pneumocystis carinii pneumonia. Ann Intern Med. 1970 Nov;73(5):761-5. doi: 10.7326/0003-4819-73-5-761. No abstract available. PMID 5312204
- [Background] Sepkowitz KA, Telzak EE, Gold JW, Bernard EM, Blum S, Carrow M, Dickmeyer M, Armstrong D. Pneumothorax in AIDS. Ann Intern Med. 1991 Mar 15;114(6):455-9. doi: 10.7326/0003-4819-114-6-455. PMID 1994791
- [Background] Coker RJ, Moss F, Peters B, McCarty M, Nieman R, Claydon E, Mitchell D, Harris JR. Pneumothorax in patients with AIDS. Respir Med. 1993 Jan;87(1):43-7. doi: 10.1016/s0954-6111(05)80312-9. PMID 8438099
- [Background] Tumbarello M, Tacconelli E, Pirronti T, Cauda R, Ortona L. Pneumothorax in HIV-infected patients: role of Pneumocystis carinii pneumonia and pulmonary tuberculosis. Eur Respir J. 1997 Jun;10(6):1332-5. doi: 10.1183/09031936.97.10061332. PMID 9192938